CLINICAL TRIAL: NCT00703989
Title: The Role of the Glucosamine Pathway and Reactive Oxygen Species in the Pathogenesis of Diabetic Complications
Brief Title: Reactive Oxygen Species in the Pathogenesis of Diabetic Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Michael Brownlee, M.D., Albert Einstein College of Medicien
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-582; JDRF grant #8-2003-784; GCRC grant # MO1-RR12248
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2008-06

CONDITIONS: Type 1 Diabetes
Keywords: hyperglycemia; diabetic complications; advanced glycation endproducts; hexosamine pathway; prostacyclin synthase; reactive oxygen species
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia; Diabetes Complications | interventions — benphothiamine; Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Patients with Type 1 diabetes
  Interventions: Dietary Supplement: benfotiamine, α-lipoic acid
- II (No Intervention): Age-matched male subjects without Type 1 diabetes

INTERVENTIONS:
Dietary Supplement: benfotiamine, α-lipoic acid — benfotiamine 300 mg twice a day, (Advanced Orthomolecular Research, Calgary, AB,CANADA) and slow-release α-lipoic acid (600 mg twice a day) (MRI, San Francisco, CA) for a total duration of four weeks
  Other Names: benfotiamine 300 mg .slow-release; α-lipoic acid (600 mg twice a day)
  Arms: I

SUMMARY:
Benfotiamine blocks three major pathways of hyperglycemic damage and prevents experimental diabetic retinopathy and incipient nephropathy in these models. In cultured vascular cells, it also reduces aldose reductase gene expression, activity, and sorbitol levels. It does so by activating the enzyme transketolase. α-lipoic acid, a potent antioxidant, has also been reported to reduce both diabetic microvascular and macrovascular complications in animal models. To determine whether benfotiamine in combination with α-lipoic acid would normalize markers of ROS-induced pathways of complications in humans, we performed a pilot study in subjects with Type 1 diabetes using one daily dose of benfotiamine in combination with α-lipoic acid.

DETAILED DESCRIPTION:
The glycemic status of study patients was assessed by measuring baseline values of HbA1c, fructosamine, and fasting plasma glucose. Mean HbA1c was 8.7+ 0.7%, mean fructosamine was 421+29 mg/dl (normal range 174-286 mg/dl), and mean fasting blood glucose was 198+44 mg/dl.

At day 0, subjects levels of markers of two benfotiamine-sensitive pathways were determined: intracellular advanced glycation endproduct (AGE) formation, as reflected by a marker of increased intracellular methylglyoxal adducts in endothelial cells, angiopoietin 2 and hexosamine pathway activity, measured by determination of N-acetylglucosamine-modified protein in circulating monocytes. PKC activity in circulating monocytes could not be measured because the amount of blood required exceeded that approved by the Committee on Clinical Investigations. Serum levels of 6-keto-PGF-1 , a stable product produced by the nonenzymatic hydration of the antiatherogenic mediator prostacyclin were also determined. Subjects then took benfotiamine 300 mg twice a day, (Advanced Orthomolecular Research, Calgary, AB,CANADA) and slow-release α-lipoic acid (600 mg twice a day) (MRI, San Francisco, CA) for 28 days. Blood was obtained at day 0, day 15, and day 28.

Data were analyzed using 1-factor analysis of variance to compare the means of all the groups. The Tukey-Kramer multiple comparisons procedure was used to determine which pairs of means were different.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Type 1 diabetes duration between zero and fifteen years
* current insulin therapy

Exclusion Criteria:

* Female
* proliferative retinopathy
* microalbuminuria
* symptomatic diabetic neuropathy
* cardiovascular disease
* taking medications
* smoking

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
intracellular advanced glycation endproducts | four weeks
hexosamine pathway | four weeks
prostacyclin synthase activity | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brownlee, M.D., Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- GCRC, Albert Einstein College of Medicine, The Bronx, New York, United States

REFERENCES:
- [Background] Brownlee M. The pathobiology of diabetic complications: a unifying mechanism. Diabetes. 2005 Jun;54(6):1615-25. doi: 10.2337/diabetes.54.6.1615. No abstract available. PMID 15919781
- [Derived] Du X, Edelstein D, Brownlee M. Oral benfotiamine plus alpha-lipoic acid normalises complication-causing pathways in type 1 diabetes. Diabetologia. 2008 Oct;51(10):1930-2. doi: 10.1007/s00125-008-1100-2. Epub 2008 Jul 29. PMID 18663426